CLINICAL TRIAL: NCT03466086
Title: Clinical Evaluation of Two Marketed Artificial Tears in Non-contact Lens Wearing Patients
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Johnson & Johnson Vision Care, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: CR-6013
Record Dates: First submitted 2018-02-26; First posted 2018-03-15 (Actual); Results first posted 2019-05-29 (Actual); Last update posted 2019-06-28 (Actual); Status verified 2019-06

CONDITIONS: Visual Acuity

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (2):
- Test/Control (Experimental): Subjects between the ages of 18-69 years of age will sequentially try the Test and Control eye drops in a random order
  Interventions: Device: Test Eye Drops; Device: Control Eye Drops
- Control/Test (Experimental): Subjects between the ages of 18-69 years of age will sequentially try the Control and Test eye drops in a random order.
  Interventions: Device: Test Eye Drops; Device: Control Eye Drops

INTERVENTIONS:
Device: Test Eye Drops — blink® intensive TRIPLE ACTION 3 in 1 eye drops
Device: Control Eye Drops — Systane® BALANCE eye drops

SUMMARY:
This clinical study is a randomized, double-masked, cross-over, bilateral, 2 treatment x 2 period, dispensing 4-visit study with a 7-9 day washout period in between visits 2 and 3. The study will last approximately 3 months.

ELIGIBILITY:
Inclusion Criteria:

* Potential subjects must satisfy all the following criteria to be enrolled in the study:

  1. Subjects must be at least 18 years of age and no more than 69 years of age (inclusive)
  2. Subjects must be non-contact lens wearers
  3. Subjects must have a DEQ-5 score of >6 at either Visit 0 (pre-screen) and/or Visit 1 (screening).
  4. Subjects must achieve visual acuity of 20/30 (equivalent to 0.18 logMAR) or better in each eye, either unaided or best corrected.
  5. Subjects must possess a functional/usable pair of spectacles and bring them to every visit (only if applicable - to the investigators discretion).
  6. Subjects must read, understand, and sign the Statement of Informed Consent.
  7. Subjects must appear able and willing to adhere to the instructions set forth in this clinical protocol

     Exclusion Criteria:
* Potential subjects who meet any of the following criteria will be excluded from participating in the study:

  1. Currently pregnant or breast-feeding.
  2. Diabetes.
  3. Any ocular or systemic allergies or disease which may interfere with the clinical trial (at the investigator's discretion).
  4. Any systemic disease, autoimmune disease, or use of medication which may interfere with the clinical trial (at the investigator's discretion).
  5. Any infectious diseases (e.g. hepatitis, tuberculosis) or a contagious immunosuppressive disease (e.g. HIV), by self-report
  6. Any Grade 3 or greater biomicroscopy findings (this includes, corneal edema, corneal staining, corneal vascularization, conjunctival injection, tarsal abnormalities, bulbar injection) on the FDA scale
  7. Any active ocular abnormalities/conditions that may interfere with the clinical trial (this includes, but not limited to, chalazia, recurrent styles, pterygium, infection, etc)
  8. Any corneal distortion due to previous rigid gas permeable lens wear, surgery or pathology
  9. History of any ocular or corneal surgery (e.g. RK, PRK, LASIK)
  10. Participation in any pharmaceutical or medical device related clinical trial within 14 days prior to study enrollment.
  11. History of binocular vision abnormality or strabismus.
  12. Habitual wearers of soft contact lenses in the past 1 month or rigid gas permeable lens within the past 3 months
  13. Current habitual use of Prescription Only Medicines (POM) to treat dry eye or ocular discomfort, ocular steroids, or any medication (RX or OTC) that would interfere with the clinical study (at the discretion of the investigator).)
  14. Employees of investigational clinic (investigator, coordinator, and technician etc) or family member of an employee of the clinical site by self-report.

In addition to the above criteria, patients with any allergy or sensitivity to ingredients that this product may contain (liposomes, sodium hyaluronate, vitamin E polyethylene glycol succinate (TPGS), polyethylene glycol 400 (PEG 400), disodium edetate, polyhexanide methylbiguanide, propylene glycol, boric acid, dimyristoyl phosphatidylglycerol, edetate disodium, hydroxypropyl guar, mineral oil, polyoxyl 40 sterate, polyquaternium-1, sorbitan tristearate, sorbitol, hydrochloric acid and/or sodium hydroxide) should not participate in the study.

Ages: 18 Years to 69 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 57 (Actual)
Dates: Start 2018-02-09 (Actual); Primary Completion 2018-05-16 (Actual); Study Completion 2018-05-16 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- The University of Manchester, Manchester, United Kingdom

RESULTS

PARTICIPANT FLOW:
Recruitment Details: A total of 57 subjects were enrolled in this study, of which 55 subjects were assigned to receive at least 1 eye drop while, 2 subjects were screen failures and/or not assigned. Of the total assigned subjects, 53 subjects completed the study and 2 subjects discontinued the study.
Groups:
- Test/Control: Subjects randomized to this sequence received the Test eye drop during the first period and then received the Control eye drop during the second period.
- Control/Test: Subjects randomized to this sequence received the Control eye drop during the first period and then received the Test eye drop during the second period.
Period: Period 1
Arm/Group | Test/Control | Control/Test
Started | 28 | 27
Completed | 26 | 27
Not Completed | 2 | 0
Not completed — Sponsor decision due to study timeline | 1 | 0
Not completed — Withdrawal by Subject | 1 | 0
Period: Period 2
Arm/Group | Test/Control | Control/Test
Started | 26 | 27
Completed | 26 | 27
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Dispensed Subjects: All subjects dispensed at least one eye drop and 1 contact lens
Arm/Group | Dispensed Subjects
Number analyzed (Participants) | 55
Age, Continuous [Mean (Standard Deviation); unit: Years] | 26.76 (11.273)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 37
  Male | 18
Race/Ethnicity, Customized [Number; unit: Participants]
  Asian | 13
  Black Or African American | 4
  White | 34
  Other | 4
Region of Enrollment [Count of Participants; unit: Participants]
  United Kingdom | 55

OUTCOME MEASURES:

1. Primary Outcome: Ocular Comfort
Description: Ocular comfort was measured using the visual analogue scale of 0 to 100. Where 0 is extremely uncomfortable and 100 is extremely comfortable.
Time Frame: 1-Week Follow-up
Population: All subjects that completed all study visits without a major protocol deviation.
Measure: Mean (Standard Deviation); unit: Units on a scale
Units Other Than Participants: eyes
Groups:
- Test: All subjects that wore the Test eye drop during either the first or second period of the study.
- Control: All subjects that wore the control eye drop in either the first or second period of the study.
Arm/Group | Test | Control
Number analyzed (Participants) | 52 | 52
Number analyzed (eyes) | 104 | 104
Units on a scale | 81.96 (12.407) | 82.49 (15.238)
Statistical Analysis 1: Comparison: Test vs Control; Test type: Superiority — This was a pilot study and the sample size was not based on any empirical power calculation; Multivariate Bayesian Model — Superiority will be declared if the lower bound of the 2-sided 95% credible interval of the difference between Test and Control is greater than 0; The correlation between measurements across periods were modeled using unstructured variance-covariance matrix; Mean Difference (Final Values) = 0.13, 95% CI 2-sided [-2.35 to 2.59], Standard Deviation 1.238 — Mean Difference was calculated as Test minus Control

2. Secondary Outcome: Subjective Dryness Rating
Description: Subjective dryness was assessed using Ocular Surface Disease Index (OSDI©) instrument. Dryness is evaluated on a scale of 0 to 100, where higher scores indicate more symptoms of dryness
Time Frame: 1-Week Follow-up
Population: All subjects that completed all study visits without a major protocol deviation.
Measure: Mean (Standard Deviation); unit: Units on a Scale
Arm/Group | Test | Control
Number analyzed (Participants) | 52 | 52
Units on a Scale | 25.68 (10.162) | 24.69 (10.609)
Statistical Analysis 1: Comparison: Test vs Control; This was a pilot study and the sample size was not based on any empirical power calculation; Test type: Superiority — Superiority will be declared if the lower bound of the 2-sided 95% credible interval of the difference between Test and Control is less than 0; Multivariate Bayesian Analysis; The correlation between measurements across periods were modeled using unstructured variance-covariance matrix; Mean Difference (Final Values) = 1.49, 95% CI 2-sided [-0.40 to 3.37], Standard Deviation 0.951; Mean difference was calculated as Test - Control

ADVERSE EVENTS:
Time Frame: Throughout the entire duration of the study. Approximately 3 week per subject.
Groups:
- Test: All subjects that wore the Test eye drop during either period 1 or period 2 during the study.
- Control: All subjects that wore the Control eye drop during either period 1 or period 2 during the study.
Arm/Group | Test | Control
All-Cause Mortality (participants affected / at risk) | 0/55 | 0/55
Serious Adverse Events (participants affected / at risk) | 0/55 | 0/55
Other Adverse Events (participants affected / at risk) | 0/55 | 0/55

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2018-01-03): https://cdn.clinicaltrials.gov/large-docs/86/NCT03466086/Prot_SAP_000.pdf